CLINICAL TRIAL: NCT05977504
Title: The Effectiveness of "Multi-Psychological Empowerment" Courses Through Remote, Digital Media, Workshop Intervention for Oncology Nurses on Physical and Psychological Status, Self-Efficacy and Communication Ability
Brief Title: The Effectiveness of "Multi-Psychological Empowerment" Courses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202302085RINC
Record Dates: First submitted 2023-07-03; First posted 2023-08-04 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Cancer; Oncology; Psychological; Self Efficacy; Communication
Keywords: Training course; Oncology nurse; Psychological support; Self-efficacy
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Psychological Empowerment Courses (Experimental): 9 times online course and 3-days workshop for 6 months .
  Interventions: Other: Multi-Psychological Empowerment Courses
- Control group (No Intervention): Participants in control group will receive usual course.

INTERVENTIONS:
Other: Multi-Psychological Empowerment Courses — 9 times online course and 3-days workshop for 6 months of psychological Empowerment Courses.
  Arms: Multi-Psychological Empowerment Courses

SUMMARY:
In the first-year project of this study, oncology nurses have reported experiencing massive stress, insufficient communication ability, and the need for communication-related training. 70% of them had moderate or higher severity of workload, fatigue, and psychological distress (at the measure point) before being provided with Basic Remote Psychological Support Course (BRPSC). A month after BRPSC, some oncology nurses have indicated/affirmed the benefits of undergoing the comprehensive psycho oncology education training courses. Thus, the second- and third-year continuation projects are focused on the development and delivery of Multi-Psychological Empowerment Courses (MPEC) for oncology nurses

ELIGIBILITY:
Intervention group

* Inclusion Criteria:
* Over 20 years old (inclusive)
* Oncology nurses currently working in clinical practice
* At least receiving one course related to oncology nurse training, such as chemotherapy for nursing staff or oncology advanced training courses.
* Exclusion Criteria:
* Those who are unwilling or unable to participate in this course training for a full one- year period.

Control group Oncology nurses who do not need to be recruited for the comparison group will be students who participated in the remote psychological support course of the first year project effective comparison groups.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The change in Physical and Psychological Symptoms | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  The change in oncology nurses' physical and psychological state will be measured by physical and psychological state survey. It use Numerical Rating Scale(VRS) 0-10. It is a 11 Point Likert Scale (e. g. 0 is no pain; 10 is unbearable pain).
The change in Workload | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  The change in oncology nurses' workload will be measured by the self-designed scale using VRS (Numerical Rating Scale). It measures the subjective perception of oncology nurses about their workload in the past week, with scores ranging from 0 to 10.The higher the score, the greater the workload of the oncology nurses.

SECONDARY OUTCOMES:
Self efficacy scale (GSES) | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  Oncology nurses' self-efficacy were measured by self efficacy scale. There are 10 questions about the level of confidence in these situations. It's a 4 point (1-4),higher the score means the more confident you have. There is also 11 point (0-10) scale that higher the score means the more confident you are in caring for patients.
Communication ability scale | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  Oncology nurses' communication skills were measured by communication ability scale.It is a 5 Liker scale(1-5),higher scores represent better communication skills.
Efferson Empathy Scale | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  Oncology nurses' empathy were measured by Efferson Empathy Scale. It is a 7 Liker scale(1-7),higher scores means someone have more empathy.
Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being （FACIT-Sp） | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  Oncology nurses' spiritual well-being were measured by FACIT-Sp.It is a 5 Liker scale(0-4),higher scores represent better well-being.
Burnout Inventory survey | 5 time points: Time 1 (before the course) ; after the course starts, Time 2: 4th weeks ; Time3: 8th weeks；Time 4:12th weeks；Time 5(back to work 1 month)
  Oncology nurses' burnout will be measured by Burnout Inventory survey.It is a 7 Liker scale(0-6),higher scores represent high level burnout .

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan